CLINICAL TRIAL: NCT01964612
Title: Illness Crisis Adapting in Early or Middle Phase of Patient With Chronic Disease: Study of Meta-cognition Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201205106RIC
Record Dates: First submitted 2013-10-08; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Drug or Chemical Induced Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Patient with chronic disease learning of a chronic illness quickly changes the way they encounter in physiological, psychological and social aspects. The investigators research purposes will use the meta-cognitive approach to explore adjustment to life-threatening illness (ex. hypertension and diabetes) of patients may find the important factors in their coping process.

DETAILED DESCRIPTION:
Patient with chronic disease learning of a chronic illness quickly changes the way they encounter in physiological, psychological and social aspects. They need adjust themselves and their crisis lives, and some plan they had made the near or distant future. The investigators research purposes will use the meta-cognitive approach to explore adjustment to life-threatening illness (ex. hypertension and diabetes) of patients may find the important factors in their coping process.Research methods will separate three year project to describe. First year project will use qualitative methods from bio-psychosocial aspects to interview participants who may suffer illness after diagnosis or stable treatment during middle phase of illness. Second year will invite diabetes and hypertension patients from different phase of illness with different levels of health anxiety trait, meta-cognitive and control strategies if derived different coping and emotions outcome. The third year will design motivational psycho-education program for patients to alleviate the emotions and use cold meta-cognition to due good health behavior and self care with their illness. The expected results will like to test the investigators new model in caring chronic disease patients.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 20 and above, with hypertension or diabetes or both diseases.

Exclusion Criteria:

* adults with other severe physical diseases.
* adults with relevant psychological diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with obvious chronic diseases of hypertension or diabetes, or both diseases diagnosed by doctors in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
self-monitoring and self-control scale | one year

SECONDARY OUTCOMES:
meta-thinking awareness scale | one year
negative self thinking scale | one year
depression and anxiety scale | one year
life change scale | one year
health anxiety scale | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bee-Horng Lue, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hopital, Taipei, Taiwan, Taiwan